CLINICAL TRIAL: NCT01430793
Title: Vitamin D Dosing and Monitoring Study
Brief Title: Determination of Effective Vitamin D Replacement and Monitoring Strategies in Vitamin D Deficiency State
Acronym: EVIREST-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Muhammad Qamar Masood, Assistant Professor, Department of Medicine, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SM100404
Record Dates: First submitted 2011-09-06; First posted 2011-09-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vitamin D 600,000 IM (Active Comparator): Vitamin D3 600,000 units will be given by intramuscular injection
  Interventions: Drug: Vitamin D3 600,000 units IM
- Vitamin D 600,000 orally (Active Comparator): Vitamin D3 600,000 units will be given orally
  Interventions: Drug: Vitamin D3 600,000 Orally
- Vitamin D 200,000 IM (Active Comparator): Vitamin D3 600,000 units will be given by intramuscular injection
  Interventions: Drug: Vitamin D3 200,000 units IM
- Vitamin D 200,000 orally (Active Comparator): Vitamin D 200,000 units will be given orally
  Interventions: Drug: Vitamin D3 200,000 Orally

INTERVENTIONS:
Drug: Vitamin D3 600,000 units IM — Vitamin D3 600,000 units will be given by Intramuscular injection and then will be repeated every 2 monthly for 2 times if vitamin D levels remain < 30 ng/ml
  Other Names: Cholecalciferol
  Arms: Vitamin D 600,000 IM
Drug: Vitamin D3 600,000 Orally — Vitamin D3 600,000 units will be given orally and then will be repeated every 2 monthly for 2 times if vitamin D levels remain < 30 ng/ml
  Other Names: Cholecalciferol
  Arms: Vitamin D 600,000 orally
Drug: Vitamin D3 200,000 units IM — Vitamin D3 200,000 units will be given by Intramuscular injection and then will be repeated every 2 monthly for 2 times if level of vitamin D remain < 30 ng/ml
  Other Names: Cholecalciferol
  Arms: Vitamin D 200,000 IM
Drug: Vitamin D3 200,000 Orally — Vitamin D3 200,000 units will be given by orally and then will be repeated every 2 monthly for 2 times if level of vitamin D remain < 30 ng/ml
  Other Names: Cholecalciferol
  Arms: Vitamin D 200,000 orally

SUMMARY:
The purpose of the study is determination of effective vitamin D replacement strategy in vitamin D deficiency states with currently available preparations in Pakistan & to determine the cost effective monitoring strategy with urinary calcium excretion serving as a surrogate marker of achievement of vitamin D sufficiency state.

The study will be conducted at the out-patient Endocrinology Clinics of the Aga Khan University Hospital, Karachi, Pakistan. All patients seen in endocrine clinics with Vitamin D level less than 20 ng and do not have any of exclusion criteria mentioned below will be eligible for recruitment in the study. The study participants will be randomly assigned into 4 groups for intervention to receive intramuscular or oral Vitamin D in 200,000 or 600,000 units as per group allocation. Each group will comprise of 25 participants.

Group 1: Vitamin D3 600,000 units IM and then every 2 monthly for 2 times if levels remain < 30 ng/ml.

Group 2: Vitamin D3 600,000 units orally and then every 2 monthly for 2 times if levels remain < 30 ng/ml.

Group 3: Vitamin D3 200,000 units IM initially and then every 2 monthly for 2 months if levels remain < 30 ng/ml.

Group 4: Vitamin D3 200,000 units orally initially and then every 2 monthly for 2 times if levels remain < 30 ng/ml.

All patients will be prescribed elemental Calcium 1 gram /day. Vitamin D levels along with the other biochemical parameter and random urine for calcium & creatinine will be checked at 00, 02, 04, 06 and 12 months.

DETAILED DESCRIPTION:
Vitamin D deficiency (VDD) has resurfaced as a significant public health problem in recent years. In Pakistan and as well in the region, VDD is very prevalent despite adequate sunshine throughout the year. Prevalence of VDD of 92% and 81% in ambulatory patients has been reported from centers in Karachi and Lahore recently. Reports previously have also demonstrated VDD from various regions of Pakistan, a study conducted at tertiary care hospital in Karachi found that 55% of healthy breast fed infants and 45% of nursing mothers had very low levels of vitamin D. Another study conducted in Hazara division found rickets as a common problem in children despite abundant sunlight.

There are several areas of controversy which has great relevance for the investigators community like what level of vitamin D should be considered as deficiency, what are the daily requirements of vitamin D and how VDD should be corrected. Generally level below 20ng/ml is considered deficient and levels between 21 and 29 ng/ml is considered relative insufficiency as depicted by intestinal calcium absorption and nadir levels of parathyroid hormone.

Determination of the daily intake required to attain adequate serum 25(OH)D concentrations are compounded by the wide variability in the dose-response curve and basal 25(OH)D concentrations.

There is no universally accepted method of correcting VDD, In US the available preparation is 50,000 units of ergocalciferol, given weekly or three times per week for total of 300,000 units. Several strategies has recently been studied, a study from southern Brazil demonstrated that a single 300 000 IU oral dose of vitamin D3 was more effective than 800 IU per day to increase serum 25(OH)D levels in elderly persons, living in a low-income housing unit.

Contrary to this comparison of the equivalent oral doses of vitamin D3 600 IU/day, 4200 IU/week and 18,000 IU/month on vitamin D status showed that daily dose was more effective than a weekly dose, and a monthly dose was the least effective.

In India a recent study evaluated the common physician practice of prescribing 1500 mcg (60 000 IU) cholecalciferol per week for 8 weeks for VDD. Twenty-eight subjects with mean 25 hydoxy vitamin D level of 13.5 nmol/l received oral supplementation of 1500 mcg cholecalciferol per week and 1g elemental Ca daily for 8 weeks. At 8 weeks the vitamin deficiency was corrected in all patients with mean the mean 25(OH)D levels of 82.4 nmol/l however at 1 year follow up all subjects were again vitamin D deficient with the mean 25(OH)D level of 24.7 nmol/l. This suggests that ongoing supplementation after initial loading is needed for sustained improvement in 25(OH)D levels vitamin D levels.

In another study from Australia, a single annual intramuscular injection of 600,000 IU cholecalciferol was administered to 50 vitamin D-deficient participants. Specimens were collected at baseline and after 4 and 12 months of therapy. Serum 25OHD3 levels were significantly higher at 4 months (114 ±35 nmol/L), and 12 months (73 ±13nmol/L) compared with baseline (32 ±8nmol/L) (P < 0.001), increasing by an average of 128% over the 12 months. The therapy was effective, with normalization of serum 25OHD levels and maintenance of a level well above 50nmol/L at 12 months.

In Pakistan oral vitamin D supplementations are available in only in combination with calcium supplement with maximum availability of 400 IU. Two depot intramuscular preparations are available one with 200,000 IU and other with 600,000 IU of vitamin D3. Regarding the 600,000 unit preparation the practices among physician are varied, common practice is to give 600,000 units intramuscularly every 03 months, some physicians prescribe a second injection after first month in cases of severe deficiency and some physicians prescribe 3 injections of Vitamin D at 2 weekly interval and then repeat in 3 months if needed. Regarding the 200,000 unit preparation, it is less commonly used, more expensive than the other preparation; however it has the advantage of using orally as well. There are no published guidelines with these mega doses of depot preparations. The effects of these mega doses have not been studied in the investigators setting and practices are based on individual experiences. The investigators strongly feel that information regarding effective correction of vitamin deficiency with currently available depot preparation is lacking and the investigators study will help in answering this very important and relevant clinical query.

The investigators second objective of the study is to find a cost effective method of monitoring adequacy of vitamin D replacement. While treatment with vitamin D is easy and inexpensive, monitoring of vitamin D levels is expensive, not widely available and assay limitations in terms of precision, accuracy and measurements of status of vitamin D.

The investigators planned to measure urinary calcium excretion as an index of adequacy of vitamin D status and to determine the correlation with vitamin D levels.

Urine calcium is a reflection of dietary intake, calcium absorption from gut, bone turnover, and renal excretion mechanisms. At steady-state excretion is usually approximately 30% of the dietary intake. The efficiency of the absorption of renal calcium and of intestinal calcium and phosphorus is increased in the presence of vitamin D. Reports show increase of intestinal calcium transport by 45 to 65% in women when 25-hydroxyvitamin D levels were increased from an average of 20 to 32 ng per milliliter (50 to 80 nmol per liter).

Calciuria estimated by the calcium/creatinine ratio tended to increase in parallel with 25 OH vitamin D levels this is mostly studied in pediatric population given vitamin D for prophylaxis of rickets. In adult patients with hypercalciuria and renal stone formation positive correlation is seen with vitamin D and urinary calcium excretion. Seasonal variation in vitamin D levels and urinary calcium excretion has also been described. Gokce C et al find significant correlation between random single voided urine calcium-to-creatinine ratio and 24-hour total calcium excretion in 67 subjects who were selected prospectively to represent a wide range of renal and parathyroid function as well as urinary calcium and phosphate loss.

The investigators expect that this simple urine test can be followed to evaluate the vitamin D sufficiency state in post vitamin D treated patients and can serve as a cost effective mean of following these patients.

Objectives:

Primary Objective:

To determine the effect of vitamin D replacement on vitamin D levels with currently available preparations in patients with vitamin D deficiency.

Secondary objective:

To determine the correlation between vitamin D levels and urinary calcium excretion in deficiency and sufficiency states.

ELIGIBILITY:
Inclusion Criteria:

* All patients with Vitamin D level less than 20 ng/dl

Exclusion Criteria:

* Patients who have received vitamin D injection in last 03 months.
* Patients with hypercalcemia (corrected calcium > 10.6 mg/dl)
* Known Malignancy.
* Known case of CLD or serum ALT > 3 times ULN
* Patients with creatinine > 2.0 mg/dl.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in vitamin D levels with specified dose and route of administration, at define intervals | 02, 04, 06 and12 months

SECONDARY OUTCOMES:
Differences in the random urinary calcium to creatinine ratio in the untreated and treated state and its correlation with vitamin D levels | 00, 02, 04, 06 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Q Masood, MBBS; FACP, Principal Investigator — Aga Khan University; Abdul Jabbar, MBBS; FRCP, Study Chair — Aga Khan University; Aysha Habib, MBBS; FCPS, Study Director — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Masood MQ, Khan A, Awan S, Dar F, Naz S, Naureen G, Saghir S, Jabbar A. COMPARISON OF VITAMIN D REPLACEMENT STRATEGIES WITH HIGH-DOSE INTRAMUSCULAR OR ORAL CHOLECALCIFEROL: A PROSPECTIVE INTERVENTION STUDY. Endocr Pract. 2015 Oct;21(10):1125-33. doi: 10.4158/EP15680.OR. Epub 2015 Jul 7. PMID 26151421